CLINICAL TRIAL: NCT06190847
Title: Oral Microbiome is Associated With the Response to Chemoradiotherapy in Initial Inoperable Patients With Esophageal Squamous Cell Cancer
Status: Recruiting | Type: Observational
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Dong Qian, dr, Anhui Provincial Hospital
Other Study IDs: 2023-KY202
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Esophageal Squamous Cell Carcinoma; Chemoradiotherapy; Initial Inoperable
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: cancer
  Interventions: Other: regular chemoradiotherapy

INTERVENTIONS:
Other: regular chemoradiotherapy — regular chemoradiotherapy

SUMMARY:
Esophageal cancer accounts for more than half of the world, seriously affecting people's health in China. 95% patients are squamous cell carcinoma. Surgery is the preferred treatment for early and middle stage esophageal cancer, but patients with clinical stage T4b or other surgical contraindications have no surgical opportunity. In recent years, radical chemoradiotherapy has played a key role in the treatment of local advanced esophageal cancer with some poor predicting biomarkers. Oral bacteria may play a pathogenic role in cancer and other chronic diseases by producing chemical carcinogens and inflammatory factors through direct metabolism. A large number of studies have also suggested that tooth loss and poor oral hygiene are closely related to upper digestive tract cancer, indicating the possible role of oral microorganisms in the occurrence and development of upper digestive tract cancer, and saliva is the main source of oral flora colonization. Therefore, it is worth further research to explore the interaction between microbial metabolism imbalance and radiotherapy in patients with esophageal cancer. In summary, we intend to conduct a prospective cohort study to explore the role of salivary microbes in radiotherapy in patients with initially inoperable patients with local advanced esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years old;

  * Eastern Cooperative Oncology Group (ECOG) 0-2;
  * Esophageal squamous cell carcinoma;
  * cT2-4aN0-3M0 (AJCC 8th) confirmed by radiological examination;
  * initial unresectable at initial diagnosis confirmed by thoracic surgeons;
  * Treatment naive;
  * No contraindications for adjuvant chemoradiotherapy;
  * Signature of inform consent.

Exclusion Criteria:

* • younger than 18 years old or older than 85 years old;

  * ECOG>2;
  * Esophageal adenocarcinoma, small-cell cancer and other pathological types;
  * cT1anyNM0, cT4banyNM0, c anyTanyNM0 confirmed by radiological examination;
  * Resectable at initial diagnosis confirmed by thoracic surgeons;
  * Previous treatment of chemotherapy, radiotherapy, and other treatment;
  * Contraindications for chemoradiotherapy;
  * No signature of inform consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: initial inoperable esophageal squamous cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 97 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
pCR | 1 month post treatment

SECONDARY OUTCOMES:
EFS | 1 to 3 years
the surgical conversion rate | 1month post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Dong Qian, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided